CLINICAL TRIAL: NCT05688436
Title: Pregnancy Outcomes in Women Exposed to Diroximel Fumarate
Brief Title: A Study to Learn More About The Safety of Diroximel Fumarate (VUMERITY®) in Participants Who Took it During Pregnancy And About the Health of Their Babies
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 272MS402
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Pregnancy; Relapsing forms of Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — diroximel fumarate; Alemtuzumab; Fingolimod Hydrochloride; Glatiramer Acetate; Interferon-beta; Natalizumab; ocrelizumab; ofatumumab; ozanimod; peginterferon beta-1a; ponesimod; siponimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diroximel Fumarate (DRF): Pregnant women with MS who were exposed to DRF.
  Interventions: Drug: Diroximel Fumarate
- Non-DRF: Pregnant women with MS who were exposed to disease-modifying therapies (DMTs) other than DRF.
  Interventions: Biological: Alemtuzumab; Drug: Fingolimod; Drug: Glatiramer acetate; Biological: Interferon beta; Biological: Natalizumab; Biological: Ocrelizumab; Biological: Ofatumumab; Drug: Ozanimod; Biological: Peginterferon beta-1a; Drug: Ponesimod; Drug: Siponimod
- Non-DMT: Pregnant women with MS who were not exposed to DMTs.

INTERVENTIONS:
Drug: Diroximel Fumarate — Administered as specified in the treatment arm.
  Other Names: VUMERITY; BIIB098
  Groups: Diroximel Fumarate (DRF)
Biological: Alemtuzumab — Administered as specified in the treatment arm.
  Groups: Non-DRF
Drug: Fingolimod — Administered as specified in the treatment arm.
  Groups: Non-DRF
Drug: Glatiramer acetate — Administered as specified in the treatment arm.
  Groups: Non-DRF
Biological: Interferon beta — Administered as specified in the treatment arm.
  Groups: Non-DRF
Biological: Natalizumab — Administered as specified in the treatment arm.
  Other Names: Tysabri; BG00002
  Groups: Non-DRF
Biological: Ocrelizumab — Administered as specified in the treatment arm.
  Groups: Non-DRF
Biological: Ofatumumab — Administered as specified in the treatment arm.
  Groups: Non-DRF
Drug: Ozanimod — Administered as specified in the treatment arm.
  Groups: Non-DRF
Biological: Peginterferon beta-1a — Administered as specified in the treatment arm.
  Groups: Non-DRF
Drug: Ponesimod — Administered as specified in the treatment arm.
  Groups: Non-DRF
Drug: Siponimod — Administered as specified in the treatment arm.
  Groups: Non-DRF

SUMMARY:
In this study, researchers will learn more about the effects of diroximel fumarate (DRF), also known as VUMERITY®, when taken during pregnancy in people with multiple sclerosis, also known as MS. In MS, the immune system attacks the nerves in the brain and spinal cord. The affected areas are called lesions. The damage makes it difficult for the brain and spinal cord to function and send messages throughout the body. MS can be a progressive disease, which means it may get worse over time. In relapsing forms of MS (RMS), new symptoms may happen, and existing symptoms may get better or worse over time. DRF is an approved drug that is used to treat people with RMS.

This is known as an "observational" study, which collects health information about study participants without changing their medical care. The main goal of this study is to collect birth and health information from 3 groups of participants and their babies. These groups are:

* Those who took DRF during their pregnancy
* Those who took other drugs for RMS during their pregnancy, but not DRF
* Those who did not take any drugs for RMS during their pregnancy

The main question researchers want to learn about in this study is:

• How many participants' babies were born with major congenital malformations (MCMs)? MCMs are problems with how a baby's body forms before birth.

Researchers will also learn more about:

* Loss of the baby before 20 weeks of pregnancy
* Loss of the baby at and after 20 weeks of pregnancy
* How many babies are born early (at or before 37 weeks)
* How many babies are small for their age while in the participant's uterus
* How many babies are born with any sign of life

This study will be done as follows:

* Participants with RMS can join this study if they become pregnant from 29th October 2019 to 31st July 2030. Information will start being collected when the participant decides to join the study.
* The participants' medical records will be reviewed 2 times during the study - once when the study is halfway done, and one at the end of the study.
* Each participant will be in the study until the end of their pregnancy. Each baby will be in the study for up to 1 year after birth.
* The study is planned to end by 30th April 2031.

DETAILED DESCRIPTION:
The primary objective of the study is to estimate the prevalence of major congenital malformations (MCMs) and compare the prevalence between the diroximel fumarate (DRF) and comparator groups. The secondary objectives of the study are to estimate the incidence of spontaneous abortion (SA) and compare the incidence between the DRF and comparator groups; to estimate the incidence of preterm birth and compare the incidence between the DRF and comparator groups; to estimate the incidence of stillbirth and compare the incidence between the DRF and comparator groups; to estimate the prevalence of small for gestational age (SGA) and compare the prevalence between the DRF and comparator groups; and to estimate the incidence of live birth and compare the incidence between the DRF and comparator groups.

ELIGIBILITY:
Key Inclusion Criteria:

* Last menstrual period (LMP) between 29 October 2019 and 31 July 2030.
* Continuous medical and pharmacy coverage for a minimum of 6 months prior to and including the estimated LMP.
* Presence of MS.

Key Exclusion Criteria:

- Pregnancies will be excluded from this study if they are exposed to any known teratogens from the beginning of baseline through the end of the relevant exposure window.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The participants included in this study will be drawn from the population of adult women with MS who become pregnant between 29 October 2019 and 31 July 2030.
Sampling Method: Non-Probability Sample
Enrollment: 1178 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2031-01-17 (Estimated); Study Completion 2031-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of Major Congenital Malformations (MCMs) | Up to 52 weeks postdelivery
  MCMs includes abnormalities in structural development that are medically or cosmetically significant are present at birth and persist in postnatal life unless or until repaired.

SECONDARY OUTCOMES:
Number of Spontaneous Abortions | Before 20 weeks of gestation
  Spontaneous abortion is defined as the loss of a fetus due to natural causes before 20th week of gestation.
Number of Preterm Births | At or before the 37 weeks of gestation
  Preterm birth is defined as a live birth at or before the 37th week of gestation.
Number of Stillbirths | At or after the 20 weeks of gestation
  Stillbirth is defined as the loss of pregnancy at or after the 20th week of gestation.
Number of Small for Gestational Age (SGA) | Up to 52 weeks postdelivery
  SGA is defined as birthweight below the 10th percentile for gestational age.
Number of Live Births | Up to delivery (approximately 10 months)
  Livebirth is defined as a delivered fetus with any sign of life (e.g., voluntary movement, heartbeat) regardless of gestational weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- OptumInsight, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/